CLINICAL TRIAL: NCT06355492
Title: Effectiveness of Virtual Reality Distraction During Infiltration Anesthesia in Pediatric Patients.
Brief Title: Virtual Reality Distraction in Pediatric Patients.
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Rokia Abdelrhman Saad Elfaramawy, Pediatric Dentistry, Oral Health and Preventive Dentistry Department, Tanta University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 2090/10/30
Record Dates: First submitted 2024-04-04; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Virtual Reality; Distraction; Infiltration Anesthesia; Pediatric Patients

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Patients will take buccal infiltration anesthesia using (regular screen).
  Interventions: Device: regular screen
- VR group (Experimental): Patients will take buccal infiltration anesthesia using (Virtual reality goggles).
  Interventions: Device: Virtual reality goggles (VR )

INTERVENTIONS:
Device: Virtual reality goggles (VR ) — Patients will take buccal infiltration anaethesia using (Virtual reality goggles) that properly adjusted around the patient's head and in front of his/her eyes.
  Arms: VR group
Device: regular screen — Patients will take buccal infiltration anaethesia using (regular screen ).
  Arms: Control group

SUMMARY:
The aim of this study is to evaluate the effect of virtual reality distraction on pain and anxiety during infiltration anesthesia in pediatric patients.

DETAILED DESCRIPTION:
Proper pain control and discomfort reduction during dental treatment, especially among children, can maximize a child's cooperation, overall satisfaction, build a good dentist-patient relationship, and enhance patient compliance. Psychological and pharmaceutical methods, and their combinations have tried to address this pain. Pharmaceutical approaches include the application of topical anesthetics. Psychological and behavioral modification methods including active distractions, deep breathing, Witaul and eye movement distractions. Passive distraction methods, such as audiovisual glasses and video distraction. Other methods, such as precooling the injection site, warming the local anesthesia, and camouflaging the syringe, have also been suggested.

A range of fear management techniques have been described in the literature and American Academy of Pediatric Dentistry (AAPD) has described some concepts as basic behavior guidance such as communication, tell show do, voice control, nonverbal communication, positive reinforcement, distraction and parental absence/presence, and advanced behavior guidance such as protective stabilization, sedation and general anesthesia.

Distraction as a behavior guidance technique is defined by the American Academy of Pediatric Dentistry (AAPD) as the technique of diverting the patient's attention from what may be perceived as an unpleasant procedure.

Audiovisual distraction techniques are used in dental clinics and have shown great results in managing anxious pediatric patients.

Virtual reality (VR) distraction, defined as a human-computer interface that enables the user to interact dynamically with the computer- generated environment is a new method in the medical field with the aim of aiding in patient behavior management. It offers the advantage of an immersive virtual experience blocking out external stimuli that may provoke a negative attitude, especially in young patients.

Distraction using VR provided favorable outcomes for adult and pediatric patients during various dental procedures, ranging from simple anesthesia to periodontal, restorative, and pulpal therapy .

ELIGIBILITY:
Inclusion Criteria:

1. Healthy children with no systemic illness.
2. Cooperative child with frankels behavior rating scale positive or definitely positive.
3. Patient requiring infiltration LA for dental treatment.
4. Children with proper parental consent.
5. Patients who needed non-urgent dental treatment.

Exclusion Criteria:

1. Medical disability such as history of seizures, convulsion disorder, vertigo, eye problems and autism.
2. Children below 5 years of age.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Assessment of pain during virtual reality distraction | After 2 weeks from the first visit.
  During local anesthesia administration, the face, legs, activity, cry, consolability (FLACC) behavioral pain assessment scale (objective scale) will be recorded to assess pain. Immediately after anesthetic administration, the patients will be placed in upright position and will be shown Wong-Baker faces pain rating scale (subjective scale) and give a brief explanation to the child about each face and instruct the child to choose the face that describe their feeling during administration of local anaethesia

CONTACTS AND LOCATIONS:
Locations (1):
- Rokia Abdelrhman Saad Elfaramawy, Tanta, El-Gharbia, Egypt

REFERENCES:
- [Background] Kamath PS. A novel distraction technique for pain management during local anesthesia administration in pediatric patients. J Clin Pediatr Dent. 2013 Fall;38(1):45-7. doi: 10.17796/jcpd.38.1.265807t236570hx7. PMID 24579282
- [Background] Custodio NB, Costa FDS, Cademartori MG, da Costa VPP, Goettems ML. Effectiveness of Virtual Reality Glasses as a Distraction for Children During Dental Care. Pediatr Dent. 2020 Mar 15;42(2):93-102. PMID 32276674
- [Background] Al-Khotani A, Bello LA, Christidis N. Effects of audiovisual distraction on children's behaviour during dental treatment: a randomized controlled clinical trial. Acta Odontol Scand. 2016 Aug;74(6):494-501. doi: 10.1080/00016357.2016.1206211. Epub 2016 Jul 13. PMID 27409593